CLINICAL TRIAL: NCT02623842
Title: Radiofrequency Non-ablation in the Treatment of Women With Urinary Stress Incontinence: Study Pilot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: U1111-1166-4522
Record Dates: First submitted 2015-12-01; First posted 2015-12-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-11

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; woman; radiofrequency
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiofrequency (Experimental)
  Interventions: Device: Tonederm® (Radiofrequency non ablative)

INTERVENTIONS:
Device: Tonederm® (Radiofrequency non ablative) — The application of RF was performed by physical therapist trained in the technique of radio frequency through the Tonederm® brand device with capacitive transfer method using non-ablative handle with electrode in the region of the external urethral meatro and coupling electrode placed on the participant's back. For application, the participants were in gynecological position. The session had an average duration of 20 minutes. The temperature was measured by an infrared thermometer when it reached 41graus radiofrequency was maintained for 2 minutes.

SUMMARY:
Pilot study, case series conducted in women with a clinical diagnosis of urinary incontinence and were treated with radiofrequency technique for capacitive transfer non ablative in external urethral meatus. All participants did an hour Pad Test. The participants made five sessions of Radio Frequency (RF) with an interval of seven days between them. The application of RF was performed by physical therapist trained in the technique of radio frequency through the Tonederm® brand device with capacitive transfer method using non-ablative handle with electrode in the region of the external urethral meatro and coupling electrode placed on the participant's back. For application, the participants were in gynecological position. The session had an average duration of 20 minutes. The temperature was measured by an infrared thermometer when it reached 41graus radiofrequency was maintained for 2 minutes.

ELIGIBILITY:
Inclusion Criteria:

* The target audience was made up of women aged between 18 and 65 years with a diagnosis of stress urinary incontinence, referred for physical therapy and who had Pad Test positive criteria by International Continence Society

Exclusion Criteria:

* Were excluded from the study participants with limited understanding, with neurological degenerative chronic diseases, sensory deficit in the genital region, users of pacemaker and intrauterine device of copper and pregnant women

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pad test 1 hour (urinary loss) | one week, one month, two month , three month and six month measure the urinary loss
  The pad test 1 hour is performed following some standard activities to mention the amount of urinary loss, through an absorbent delivered the patients ... after the completion of the activities the absorbent is heavy.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia V Lordelo, PhD, Principal Investigator — Centro de Atenção ao Assoalho Pélvico - BAHIANA